CLINICAL TRIAL: NCT04312659
Title: A Multi-Center Registry Study of Infliximab in the Treatment of Chinese Children With Crohn's Disease
Brief Title: A Study of Infliximab in the Treatment of Chinese Children With Crohn's Disease
Status: Completed | Type: Observational
Sponsor: Johnson & Johnson (China) Investment Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR108748; C0168CRD4020 (Other: Johnson & Johnson (China) Investment Ltd.)
Record Dates: First submitted 2020-03-03; First posted 2020-03-18 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease | interventions — Infliximab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Infliximab: Participants with pediatric Crohn's disease (CD) who were treated with Infliximab (IFX) and signed the Informed Consent Form (ICF) for the study will be enrolled case by case. Each participants will be followed up for at least 30 weeks. After 30 weeks, participants continuing IFX treatment will be followed up, with a maximum follow-up period of 102 weeks. The primary data source will be participants medical records for all data entered into the CRF.
  Interventions: Drug: Infliximab

INTERVENTIONS:
Drug: Infliximab — Participants will be observed who were treated with Infliximab.

SUMMARY:
The main purpose of this study is to record the use of Infliximab (IFX) in the treatment of Chinese children with Crohn's disease (CD) in routine clinical practice and to summarize the clinical efficacy and safety of IFX in the treatment of pediatric CD.

ELIGIBILITY:
Inclusion Criteria:

* Must have a confirmed diagnosis of Crohn's disease
* Must sign, and their legal guardians/legally-acceptable representative where applicable must sign, a participation agreement/ICF allowing data collection and source data verification in accordance with local requirements
* First-time received IFX treatment

Exclusion Criteria:

* History of medical contraindications for Infliximab (IFX), example. serious infections, active tuberculosis (TB), lymphoma and other malignancies, moderate to severe heart failure, hypersensitivity to inactive components of the product or to any murine proteins
* Previous exposure to Infliximab or any other biologics
* Received an investigational drug (including investigational vaccines) or used an invasive investigational medical device within 90 days before the start of the study or the first data collection time point
* Currently enrolled in an investigational study
* Have other Crohn's-like disease that are associated with mono-genetic immune disorders

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Participants observed in this study will be pediatric participants with Crohn's disease who have signed the ICF and are treated with infliximab.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2023-09-12 (Actual); Study Completion 2023-09-12 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Clinical Response at Week 14 | Week 14
  Percentage of participants with clinical response at week 14 will be reported. Clinical response is defined as a decrease of PCDAI >=15 and total PCDAI <=30.
Number of Participants with Adverse Events (AE) as a Measure of Safety and Tolerability | Up to 102 weeks
  An AE is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.

SECONDARY OUTCOMES:
Percentage of Participants with Clinical Remission at Week 14 | Week 14
  Percentage of participants with clinical remission at week 14 will be reported. Clinical remission is defined as the total PCDAI <=10.
Percentage of Participants with Clinical Remission at Week 30 | Week 30
  Percentage of participants with clinical remission at week 30 will be reported. Clinical remission is defined as the total PCDAI <=10.
Percentage of Participants with Clinical Response at Week 30 | Week 30
  Percentage of participants with clinical response at week 30 will be reported. Clinical response defined as a decrease of PCDAI >=15 and total PCDAI<=30.
Percentage of Participants with Endoscopic Remission at Week 30 | Week 30
  Percentage of participants with endoscopic remission at week 30 will be reported. Endoscopic remission is defined as a total simple endoscopic sore for CD (SES-CD) 0-2. SES-CD is an endoscopic scoring system for CD. It is based on the score of 0-3 of the following four endoscopic variables: ulcer size, ulcerated and affected surfaces, and stenosis determined in five ileocolonic segment.
Change from Baseline in Height Z-Scores at Week 30 | Baseline and Week 30
  Change from baseline in height Z-score will be recorded directly into an electronic device and will be considered source data. Height will be measured in meters.
Change from Baseline in Body Mass Index (BMI) Z-Scores at Week 30 | Baseline and Week 30
  Change from baseline in BMI Z-score (growth and development) will be recorded directly into an electronic device and will be considered source data. BMI will be calculated based on weight (kilograms)/height (meters square).
Change from Baseline in Acute Response Indicators at Week 14 | Baseline and Week 14
  Change from baseline in acute response indicators (C response protein and erythrocyte sedimentation rate) at week 14 will be reported.
Change from Baseline in White Blood Cells Countat Week 14 | Baseline and Week 14
  Change from baseline in white blood cells count (giga cells per liter) at week 14 and will be reported.
Change from Baseline in Hemoglobin Levels at Week 14 | Baseline and Week 14
  Change from baseline in hemoglobin levels (grams per liter) will be reported at week 14.
Change from Baseline in Platelet Count at Week 14 | Baseline and Week 14
  Change from baseline in platelet count (giga cells per liter) will be reported at week 14.
Change from Baseline in Albumin Levels at Week 14 | Baseline and Week 14
  Change from baseline in albumin levels (grams per liters) will be reported at week 14.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson (China) Investment Ltd. Clinical Trial, Study Director — Johnson & Johnson (China) Investment Ltd.
Locations (5):
- China (5):
  - Guangzhou Women And Children's Medical Center, Guangzhou
  - The Childrens Hospital Zhejiang University School Of Medicine, Hangzhou
  - Ruijin Hospital Shanghai Jiao Tong University, Shanghai
  - Children's Hospital of Fudan University, Shanghai
  - Henan Children's Hospital, Zhengzhou Children's Hospital, Zhengzhou